CLINICAL TRIAL: NCT06034379
Title: Kubota Corrective Spectacles and Low Dose Atropine for Slowing Myopic Progression in Taiwanese Children
Brief Title: Electronic Spectacles Versus Low Dose Atropine in Young Myopes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Collaborators: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP1:73200-TW
Record Dates: First submitted 2023-08-26; First posted 2023-09-13 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clinical prototype (CP1) device (Experimental): 15 subjects will be randomly assigned to use the eSpectacle Clinical Prototype (CP1) device 2 hours per day, at least 6 days per week. Standard single vision correction will be used during other waking hours. The eSpectacle clinical prototype (CP1) device consists of a clear 15° central aperture and projects +9.00D defocused micro-LED lights onto the peripheral retina.
  Interventions: Device: eSpectacle Clinical prototype (CP1) device
- CP1 and 0.01% atropine (Experimental): 15 subjects will be randomly assigned to use the eSpectacle Clinical Prototype (CP1) device 2 hours per day, at least 6 days per week, in addition to nightly instillation of one drop of 0.01% atropine. Standard single vision correction will be used during other waking hours. The eSpectacle clinical prototype (CP1) device consists of a clear 15° central aperture and projects +9.00D defocused micro-LED lights onto the peripheral retina. Atropine is an anticholinergic medication which can be used for dilation and cycloplegia and has been evaluated for slowing the progression of myopia.
  Interventions: Device: eSpectacle Clinical prototype (CP1) device; Drug: 0.01% atropine
- 0.01% atropine (Experimental): 15 subjects will be randomly assigned to nightly instillation of one drop of 0.01% atropine without use of the eSpectacle clinical prototype (CP1) device. Standard single vision correction will be used during waking hours. Atropine is an anticholinergic medication which can be used for dilation and cycloplegia and has been evaluated for slowing the progression of myopia.
  Interventions: Drug: 0.01% atropine

INTERVENTIONS:
Device: eSpectacle Clinical prototype (CP1) device — The CP1 device consists of a clear 15° central aperture and projects +9.00D defocused micro-LED lights of approximately 4800 nits illumination to the peripheral retina.
  Arms: CP1 and 0.01% atropine; Clinical prototype (CP1) device
Drug: 0.01% atropine — Atropine is a and anticholinergic medication which can be used for dilation and cycloplegia.
  Arms: 0.01% atropine; CP1 and 0.01% atropine

SUMMARY:
This is a bilateral, dispensing, masked, randomized clinical trial. Myopic children will be randomly assigned to one of the following: (1) Investigational clinical prototype (CP1) device without atropine, (2) Investigational CP1 device with daily instillation of 0.01% atropine, or (3) daily instillation of 0.01% atropine without use of the investigational CP1 device. Primary endpoint: Difference in the 12-month change of cycloplegic spherical refractive error and axial length between each of the three treatment groups.

DETAILED DESCRIPTION:
The eSpectacle clinical prototype (CP1) device consists of a clear 15° central aperture and projects +9.00D defocused micro-LED lights onto the peripheral retina. In this pilot investigation, we aim to observe the ocular biometric and refractive changes following part-time wear of the clinical prototype device over a course of 12 months.

This trial is bilateral, dispensing, masked, and randomized (stratified by age). Myopic children will be randomly assigned to one of the following: (1) CP1 device without atropine, (2) CP1 device with daily instillation of 0.01% atropine, or (3) daily instillation of 0.01% atropine without use of the CP1 device.

A total of 45 subjects (15 per subgroup) are targeted to complete the study, which will consist of 8 visits: Screening, baseline/dispense, 1 week, 1 month, 3 months, 6 months, 9 months, and 12 months. Subjects will be enrolled from the patient population at the investigator site.

The primary objective is to evaluate the effectiveness of the eSpectacle clinical prototype device with and without the use of 0.01 percent atropine for slowing the progression of myopia in Taiwanese children, by assessing changes in central axial length and cycloplegic autorefraction following at least 12 hours per week of wear over 12 months. To minimize bias, the primary outcome variables of cycloplegic autorefraction and axial length will be measured by a Masked Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be between 6 and 13 years of age (inclusive).
2. The subject must appear able and willing to adhere to the instructions set forth in the clinical protocol.
3. The guardian of a minor under 18 years old must read and sign the STATEMENT OF INFORMED CONSENT and be provided a copy of the form. The subject under 18 years old must be willing to assent to the STATEMENT OF INFORMED CONSENT.
4. Spherical component of refraction in the range of -0.50 to -10.00 DS in each eye.
5. Refractive cylinder less than or equal to 2.00 DC in each eye (minus cylinder format).
6. Best corrected distance VA of at least 20/25 in each eye.

Exclusion Criteria:

1. Currently pregnant or lactating
2. History of severe dry eye, strabismus, or amblyopia
3. Any systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g., diabetes, rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with the participation in the study at the investigator's discretion.
4. Use of systemic or ocular medications (e.g., chronic steroid use) that are known to interfere with vision and ocular accommodation at the investigator's discretion.
5. Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, strabismus surgery etc.) or orthokeratology
6. Any active ocular infection.
7. Any accommodative or binocular anomalies including amblyopia.
8. Any physical or mental developmental delay.
9. Any relevant ocular or systemic condition deemed unacceptable by the investigator that may negatively impact the subject's performance or ability to successfully complete the study (at the investigator's discretion)
10. Anisometropia greater than 1.50D

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
CSER | 12 months
  Difference in the changes of cycloplegic spherical refractive error between each of the three treatment groups.
AL | 12 months
  Difference in the changes of axial length between each of the three treatment groups.

CONTACTS AND LOCATIONS:
Locations (1):
- CMU Hsinchu Hospital, Hsinchu, Taiwan